CLINICAL TRIAL: NCT06053177
Title: Primary Care Screening to Rapidly Detect Multi-organ Complications for People With Prediabetes and Type 2 Diabetes
Brief Title: Multi-morbidity Screening in People With Type 2 Diabetes and Pre Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: UoL001691
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Pre Diabetes; Obstructive Sleep Apnea; Non-Alcoholic Fatty Liver Disease; Heart Failure
Keywords: screening; multi-morbidity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Sleep Apnea, Obstructive; Non-alcoholic Fatty Liver Disease; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: Participants with type 2 diabetes
- Pre Diabetes: Participants who's most recent HbA1c is in the prediabetes range.

SUMMARY:
People with type 2 diabetes are at risk of complications linked with high blood sugars and these are monitored for in healthcare appointments. However, people with type 2 diabetes commonly suffer with additional health conditions that can affect the liver, heart and their breathing while sleeping. These conditions are thought to be caused by a similar underlying process that causes type 2 diabetes, as a result they are very common in people type 2 diabetes. Despite this they are not part of the routine health check for these people. Worryingly, current research suggests that the risk for developing these health problems, and direct complications of type 2 diabetes, can start at blood sugar levels below the threshold of type 2 diabetes. In a group of people said to have prediabetes. These people do not currently undergo annual healthcare appointments to monitor for these health complications or other linked health conditions.

This study aims to pilot a new style of clinic to address these issues. The investigators will perform a multi-morbidity assessment, where they will look for several different health problems at the same time. The investigators will be looking at health problems linked with high blood sugars, this will include problems with the liver, heart, nerves, eyes, and participants breathing overnight. They have developed a clinic visit which uses questionnaires, simple examination techniques and modern devices to try and identify these health problems.

An important part of healthcare is the burden it places on people with health problems, with this in mind the investigators will be giving the people involved in their study a voice to try and direct future research and healthcare, the investigators will ask them to provide feedback on their experience in taking part in the study and what their thoughts are in undergoing a longer but more comprehensive health appointment.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes study group

* Participants with a documented diagnosis of type 2 diabetes or HbA1c ≥48mmol/mol.
* Age ≥18 years

Prediabetes study group

* HbA1c 42 - 47 mmol/mol (inclusive) or enrolled in the diabetes prevention programme.
* Age ≥18 years

Exclusion Criteria:

* Type 1, 3 or Maturity onset diabetes of the young.
* Participants who are pregnant at the time of screening
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who are able to give their written consent and have a diagnosis of type 2 diabetes or who's latest HbA1c is ≥42mmol/mol. Who receive their medical care in the Liverpool area (UK).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2028-02-03 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
The prevalence of undiagnosed fatty liver disease with evidence of fibrosis, obstructive sleep apnoea and heart failure in people with type 2 diabetes and prediabetes | The majority of the data for this outcome measure is collected in a single study visit lasting approximatley 2 and a half hours. All data for this outcome would be collected within 4 weeks of participant enrollment.
  Participants will complete two screening questionnaires for sleep apnoea, those identified as high risk for the condition will be given a home sleep study device to confirm or reject the diagnosis. All participants will have a fibroscan to look for the presence of fatty liver disease. Participants will be screened for heart failure, with those identified as high risk undergoing an echocardiogram to confirm or reject the diagnosis.

SECONDARY OUTCOMES:
Peripheral neuropathy and cardiac autonomic dysfunction | The data for this outcome measure is collected in a single study visit lasting approximately 2 and a half hours.
  The prevalence of peripheral neuropathy and cardiac autonomic dysfunction will be assessed using specifically designed, validated and non-invasive medical devices with results compared against outcomes of the clinical peripheral neuropathy assessments (including the MNSI, painDETECT and neuropathy symptom profile questionnaires).
Multi-morbidity screening | The data for this outcome is collected as part of the primary study visit lasting approximately 2 and a half hours.
  Exploration, through a questionnaire (mixture of open ended, closed and likert questions), of participants thoughts on multi-morbidity screening in high risk groups.

CONTACTS AND LOCATIONS:
Overall Officials: Uazman Alam, PhD, Principal Investigator — The University of Liverpool
Locations (1):
- Clinical Science Centre, Aintree University Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No